CLINICAL TRIAL: NCT03767907
Title: Online Cognitive Behavioural Therapy for Addiction: Efficacy and Cost-Effectiveness in a Pragmatic Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Lena Quilty, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 073/2018
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Substance Dependence
Keywords: cognitive behavioural therapy; online treatment
MeSH Terms: conditions — Substance-Related Disorders | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Cognitive Behavioural Therapy (Experimental): Computer-based training for cognitive behavioural therapy (CBT4CBT) consists of seven modules, and includes a series of interactive videos presenting characters portrayed by professional actors struggling with real-life situations. These characters first experience a common risky situation or problem and then demonstrate the application of a targeted skill. The program further comprises games and interactive exercises to teach and model effective use of skills and strategies.
  Interventions: Behavioral: Computer-based Training for Cognitive Behavioural Therapy
- Treatment as Usual (Active Comparator): Treatment as usual consists of weekly group and/or individual psychotherapy as determined by the clinical team. Psychotherapy will include structured relapse prevention, include cognitive and behavioural techniques, motivational enhancement, mindfulness, and specialized topics (e.g., vocational training, rainbow services) as appropriate.
  Interventions: Behavioral: Treatment As Usual

INTERVENTIONS:
Behavioral: Computer-based Training for Cognitive Behavioural Therapy — Interactive content organized into seven modules, illustrating real-life scenarios associated with common risky situations, which illustrate the application of targeted skills and strategies
  Other Names: CBT4CBT
  Arms: Online Cognitive Behavioural Therapy
Behavioral: Treatment As Usual — Treatment as usual will include standard psychosocial care determined to be appropriate or necessary, on an individual patient basis.
  Arms: Treatment as Usual

SUMMARY:
The purpose of this study is to compare the efficacy and cost-effectiveness of a Computer-based Training for Cognitive Behavioural Therapy (CBT4CBT) to treatment as usual in outpatients seeking treatment for substance use disorder.

DETAILED DESCRIPTION:
Fifty-two adult outpatients seeking treatment for substance use disorder from the Centre for Addiction and Mental Health Addictions Program will be randomized to receive either a computer-based training for cognitive behavioural therapy or treatment as usual for eight weeks. Participants will complete interviews, questionnaires, and other assessments (urine toxicology and physiological assessments) at week 0, at week 8, and at 6 month follow-up). Measures will assess alcohol and drug consumption, substance use disorder symptoms and associated features, quality of life, and healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Fluency in English
3. Understanding and willingness to comply with study requirements
4. Meet diagnostic criteria for current substance use disorder
5. Have used substance in the past 30 days
6. Treatment-seeking for substance misuse

Exclusion Criteria:

1. Unable to read at sixth grade level
2. Untreated or unstable severe psychiatric or medical disorder
3. Acute suicidal or homicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Timeline Follow-Back (TLFB) | 30 days
  Frequency (days) of substance use over the past 30 days

SECONDARY OUTCOMES:
Urine Toxicology Screen | 30 days
  Determine substance use in past 30 days
Addiction Severity Index (ASI) | 30 days
  Substance Use Disorder symptom severity
  Subscale scores are calculated for 7 domains (medical, employment/support status, alcohol, drug, legal, family/social and psychological). Subscale scores are summed scores ranging from 0-1 with higher scores indicating greater problem severity.
WHO Quality of Life (WHOQOL-BREF) | 4 weeks
  Quality of Life
  Subscale scores are calculated for 4 domains (physical health, psychological, social relationships and environment) and for "overall" and "general health" quality of life. Subscale scores have a range of 0 to 100 with higher scores indicating greater quality of life.
Program and Client Costs-Substance Abuse Treatment (PACC-SAT) | 7 days
  Healthcare Costs

CONTACTS AND LOCATIONS:
Overall Officials: Lena C. Quilty, PhD, Principal Investigator — Campbell Family Mental Health Research Institute, CAMH
Locations (1):
- Campbell Family Mental Health Research Institute, CAMH, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patel A, Corman M, de Oliveira C, Mason J, Some N, Downie D, Jain E, Patterson M, Cunningham JA, George TP, Le Foll B, Quilty LC. Computer-Based Training for Cognitive Behavioural Therapy for Substance Use Disorder: A Randomized Controlled Trial Including Quantitative and Qualitative Health and Economic Outcomes: Formation informatisee pour la therapie cognitivo-comportementale pour les troubles lies a l'usage de substances : un essai randomise controle y compris les resultats quantitatifs et qualitatifs en matiere de sante et d'economie. Can J Psychiatry. 2025 Jan;70(1):9-20. doi: 10.1177/07067437241255100. Epub 2024 May 24. PMID 38783836
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.ca/research